CLINICAL TRIAL: NCT03443193
Title: The Effects of Periodization Training on Physiological Parameters, Cerebral Oxygenation, Cognitive Functions and Cardiac Remodelling in Coronary Patients.
Brief Title: Periodization of Exercise Training in Patients With Coronary Heart Disease.
Acronym: PERIOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MontrealHI 2015-1895
Record Dates: First submitted 2018-01-22; First posted 2018-02-23 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Coronary Heart Disease; Healthy Control
Keywords: aerobic exercise training; periodization; cerebral oxygenation and perfusion; cognition
MeSH Terms: conditions — Coronary Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear training (Experimental): Linear training consists to a progressive improvement of the training load during the 3 month-program.
  Interventions: Other: Exercise training
- Non-linear training (Experimental): Non-linear training consists to an undulating progressive improvement of the training load during the 3 month-program.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Patients will undergo three weekly exercise training sessions with periodized high-intensity interval training and resistance training for a period of 12 weeks.

SUMMARY:
The research project includes two components that assess exercise physiology parameters, cerebrovascular reserve, cognitive functions and cardiac function in coronary heart disease patients at rest, during an acute exercise, and after two different periodized training programs.

ELIGIBILITY:
Inclusion Criteria for patients with coronary heart disease:

* Major
* Adequate physical and mental capacities
* Autonomy in daily activities
* Documented coronary artery disease
* Stable or recent coronary artery disease

Exclusion Criteria for patients with coronary heart disease:

* Inability to complete the consent form
* Acute coronary syndrome < 3 months
* Heart failure
* Ejection fraction of the left ventricle <40%
* Coronary artery disease non revascularisable including left main coronary stenosis
* Waiting for a bridging of the coronary artery
* Chronic atrial fibrillation
* Malignant arrhythmias during exercise
* Restriction to non cardiopulmonary exercise
* Severe intolerance to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2peak) with gas exchange | At baseline and following 12 weeks exercise training intervention
  VO2peak will be measured during maximal exercise test with a gas exchange device. The highest value reached during the exercise phase of the maximal test (ergocycle) will be considered as the VO2peak. We will measure change of VO2peak before and after exercise training.

SECONDARY OUTCOMES:
Cerebral hemodynamics | At baseline and following 12 weeks exercise training intervention
  Cerebral hemodynamics will be measured using near-infrared spectroscopy (NIRS) system during maximal and submaximal exercise tests. We will measure change of cerebral hemodynamics before and after exercise training
Cognitive functions at rest by a by standard pen-paper battery test | At baseline and following 12 weeks exercise training intervention
  Cognitive functions will be measured at rest with a pen-paper battery test by a neuropsychologist. We will measure change of score to the cognitive tests before and after exercise training.
Cardiac hemodynamics | At baseline and following 12 weeks exercise training intervention
  Cardiac hemodynamics will be measured continuously during the maximal exercise test on bike using an impedance cardiography device. We will measure change of cardiac hemodynamics before and after exercise training.
Standard echocardiographic parameter of left and right ventricular strain | At baseline and following 12 weeks exercise training intervention
  global longitudinal strain (%) will be measued at rest for both ventricule

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular prevention and rehabilitation center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boidin M, David LP, Trachsel LD, Gayda M, Tremblay J, Lalonge J, Juneau M, Nigam A, Henri C. Impact of 2 different aerobic periodization training protocols on left ventricular function in patients with stable coronary artery disease: an exploratory study. Appl Physiol Nutr Metab. 2021 May;46(5):436-442. doi: 10.1139/apnm-2020-0423. Epub 2020 Oct 27. PMID 33108743
- [Derived] Trachsel LD, Boidin M, Henri C, Fortier A, Lalonge J, Juneau M, Nigam A, Gayda M. Women and men with coronary heart disease respond similarly to different aerobic exercise training modalities: a pooled analysis of prospective randomized trials. Appl Physiol Nutr Metab. 2021 May;46(5):417-425. doi: 10.1139/apnm-2020-0650. Epub 2020 Oct 23. PMID 33096006